CLINICAL TRIAL: NCT04296227
Title: Multiparameter Monitor Non-Invasive Blood Pressure Validation Study
Brief Title: Comparison of Non-Invasive Blood Pressure Methods
Acronym: NIBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vital USA, Inc. (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PR2019-329
Record Dates: First submitted 2020-02-21; First posted 2020-03-05 (Actual); Results first posted 2020-05-05 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Blood Pressure
Keywords: Blood pressure, Non-Invasive

STUDY DESIGN:
Intervention Model Description: The Vital Detect blood pressure monitor will be evaluated as a comparative, single center, non-randomized, study in a minimum of 30 subjects, conducted in 2 phases. The maximum number of subjects enrolled is 150 for both phases, to achieve 85 valid data sets. Each subject test is expected to take up to 1 hour
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ISO 81060-2:2018. (Experimental): The intended purpose of the test is to evaluate the Vital Detect blood pressure monitor to ISO 81060-2:2018. The intended use for these products are manual and automatic Non-Invasive Blood Pressure monitoring on adults age 18 and older.
  Interventions: Device: The Vital Detect blood pressure monitor

INTERVENTIONS:
Device: The Vital Detect blood pressure monitor — The end goal is to provide Non-invasive Blood Pressure (NIBP) accuracy data to support validation of the Vital Detect blood pressure monitor.

SUMMARY:
The primary objective of the study is to demonstrate the accuracy in healthy adults with Vital USA Device by comparison to a non-invasive (auscultatory) reference sphygmomanometer.

The procedure, data collection methods and data analysis that are outlined in the protocol follow the standard: International Standards Organization (ISO) 81060-2:2018 Non-invasive Sphygmomanometers - Part 2: Clinical validation of automated measurement type.

DETAILED DESCRIPTION:
This study will include up to 100 adults ≥ 18 years of age. The final subject database will contain no fewer than 85 subjects with a minimum of 255 paired observations. At least 90% of the subjects will contribute 3 paired observations, if necessary the balance of the data will be added from additional subjects.

An interim analysis will be conducted at the end of Part 1 data collection and will consist of simple statistics that will compare the test device tot he reference cuff non-invasive (auscultatory) reference sphygmomanometer.

Part 2 data collection will be conducted after Part 1 data collection interim report is reviewed and additional data collection is approved by the client. It will test an additional 55 subjects (plus extra subjects as replacements if necessary).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to provide an informed consent or have legally authorized representative consent to participate.
* Subject must be willing and able to comply with the study procedures.
* Subject must be ≥ 18
* Subject or legally authorized representative must be able to read or write in English.
* Subjects with a finger circumference < 8.3 cm.in the range of 10-25 mm
* At least 30% of subjects shall be male and at least 30% of subjects shall be female

Exclusion Criteria:

* Lack of Informed consent.
* Subjects with deformities or abnormalities that may prevent proper application of the device under test.
* Subject is evaluated by the investigator or clinician and found to be medically unsuitable for participation in this study.
* Subjects with known heart dysrhythmias
* Subjects with compromised circulation or peripheral vascular disease.
* Subjects with clotting disorders or taking prescribed blood thinners.
* Subjects that cannot tolerate sitting for up to 1 hour.
* Subject with a blood pressure demographic that has already been filled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Batchelder, Principal Investigator — Clinimark Laboratory Services; Dena M Raley, Study Director — Clinimark Laboratory Services
Locations (1):
- Clinimark Laboratory Services, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bickler PE, Schapera A, Bainton CR. Acute radial nerve injury from use of an automatic blood pressure monitor. Anesthesiology. 1990 Jul;73(1):186-8. doi: 10.1097/00000542-199007000-00030. No abstract available. PMID 2360731
- [Background] Tollner U, Bechinger D, Pohlandt F. Radial nerve palsy in a premature infant following long-term measurement of blood pressure. J Pediatr. 1980 May;96(5):921-2. doi: 10.1016/s0022-3476(80)80582-8. No abstract available. PMID 7365605
- [Background] Celoria G, Dawson JA, Teres D. Compartment syndrome in a patient monitored with an automated blood pressure cuff. J Clin Monit. 1987 Apr;3(2):139-41. doi: 10.1007/BF00858363. PMID 3585434
- [Result] Bause GS, Weintraub AC, Tanner GE. Skin avulsion during oscillometry. J Clin Monit. 1986 Oct;2(4):262-3. doi: 10.1007/BF02851174. PMID 3783197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The final study population consisted of 85 qualified healthy subjects ranging from 18 to 81 years of age of any racial / ethnic background.
Pre-assignment Details: The subjects understood the study and provided consent for participation by signing the Independent Review Board (IRB) approved Informed Consent Form prior to start of the test. The subjects were informed about the clinical investigation within his/her ability to understand following the established informed consent process.
Period: Overall Study
Arm/Group | ISO 81060-2:2018.
Started | 85
Completed | 85
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 96 six subjects were screened for this study. One subject was not enrolled, and 10 subjects were withdrawn. The final study population consisted of 85 qualified healthy subjects ranging from 18 to 81 years of age of any racial / ethnic background.
Arm/Group | ISO 81060-2:2018.
Number analyzed (Participants) | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 85
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Local subjects, within the region of Avista Adventist Hospital Plaza in Louisville, CO USA
  Participants
    United States | 85
Noninvasive Blood Pressure Measurement [Number; unit: participants] | 85

OUTCOME MEASURES:

1. Primary Outcome: Validate Non-invasive Blood Pressure Measurement Accuracy for the Vital Detect Blood Pressure Monitor.
Description: The primary objective of this study is to provide a validation for non-invasive blood pressure measurement accuracy for the Vital Detect blood pressure monitor when compared to the Reference Sphygmomanometer. Data taken was based on dual observers (Criterion 1(C1), Criterion 2 (C2) for both Systolic and Diastolic determinations. Since the same arm sequential method was used, data for a given subject were averaged to create the reference blood pressure determination against the acceptance criteria. The device under test (DUT) passed or failed the determination based on the mean error and standard deviation of the determination. The acceptance criteria:
  Criterion 1:
  Mean Error Standard Deviation (Systolic / Diastolic) (Systolic / Diastolic) </= 5.0 mmHg </= 8.0 mmHg
  Criterion 2:
  Standard Deviation (Systolic) (Diastolic) </= 5.33 mmHg </= 6.09 mmHg
Time Frame: 1 Hour
Population: The final study population consisted of 85 qualified healthy subjects ranging from 18 to 81 years of age of any racial / ethnic background. The subjects were healthy showing no evidence
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ISO 81060-2:2018.
Number analyzed (Participants) | 85
mmHg
  Systolic Pressure C1 | 4.40 (10.97)
  Systolic Pressure C2 | 4.40 (9.24)
  Diastolic Pressure C1 | 3.26 (7.21)
  Diastolic Pressure C2 | 3.26 (6.72)

ADVERSE EVENTS:
Time Frame: up to 15 days.
Arm/Group | ISO 81060-2:2018.
All-Cause Mortality (participants affected / at risk) | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85
Other Adverse Events (participants affected / at risk) | 0/85

LIMITATIONS AND CAVEATS:
Two types of device deficiencies. First was the device would go through its measurement process as expected but did not provide a reading at end of deflation.Second involved connectivity issues between the Vital Detect and the Vital USA app.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT04296227/Prot_SAP_000.pdf